CLINICAL TRIAL: NCT02650206
Title: Effect of Liraglutide on Macrophage Polarization in Human Adipose Tissue and Peripheral Blood
Brief Title: Effect of Liraglutide (Victoza) on Inflammation in Human Adipose Tissue and Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Associate Professor of Medicine; Division of Endocrinology and Metabolism, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 31063
Record Dates: First submitted 2015-06-05; First posted 2016-01-08 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type II; Diabetes Mellitus, Adult-Onset; Inflammation
Keywords: diabetes; macrophage; inflammation; adipose tissue; weight loss; liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Diabetes Mellitus; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide group (Experimental): Drug with diet control intervention: Subjects assigned to this group receive blinded pens containing liraglutide (commonly known as Victoza), manufactured by Novo Nordisk. Subjects will inject 0.6 mg daily into abdomen during the first week of the study, and if tolerated, will increase dose to 1.2 mg the second week of the study, and then up to 1.8 mg daily from the third week until the end of the 12-week study. Any adverse symptoms as well as fasting blood glucose will be monitored weekly for safety.
  Subjects, with the guidance of the study's dietitian, will remain weight-stable for the first four weeks of the study, and then will be allowed to lose weight for the remaining eight weeks of the study.
  Interventions: Drug: Victoza (liraglutide) with dietician monitoring
- Placebo group (Placebo Comparator): Diet control-only intervention: Subjects assigned to this group receive blinded pens containing placebo (normal saline) instead of liraglutide (commonly known as Victoza). Subjects will inject 0.6 mg of placebo daily during the first week of the study, will increase to 1.2 mg the second week of the study, and then up to 1.8 mg daily from the third week until the end of the 12-week study. Any adverse symptoms as well as fasting blood glucose will be monitored weekly for safety.
  Subjects, with the guidance of the study's dietitian, will remain weight-stable for the first four weeks of the study, and then will be allowed to lose weight for the remaining eight weeks of the study.
  Interventions: Other: Placebo with dietician monitoring

INTERVENTIONS:
Drug: Victoza (liraglutide) with dietician monitoring — Victoza (liraglutide), an FDA-approved medication, is a glucagon-like peptide-1 (GLP-1) receptor agonist indicated as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus. Subjects with this intervention will be followed by the MD and dietician throughout the study to monitor progress through 4 week period of weight maintenance and 8 week period of weight loss.
  Other Names: liraglutide
  Arms: Liraglutide group
Other: Placebo with dietician monitoring — Subjects will not receive the study drug, but will be followed by the MD and dietician throughout the study to monitor progress through 4 week period of weight maintenance and 8 week period of weight loss.
  Arms: Placebo group

SUMMARY:
The objective of this study is to test the hypothesis that liraglutide (commonly known as Victoza) can promote an anti-inflammatory macrophage phenotype in human adipose tissue and blood, thereby reducing localized and systemic inflammation which are risk factors for cardiovascular disease and may contribute to hyperglycemia. This will be done after 4 weeks of treatment during which weight will remain stable, and again after 12 weeks, during which liraglutide-related weight loss occurs.

DETAILED DESCRIPTION:
It has now been established that the high risk of cardiovascular disease that is associated with obesity and type 2 diabetes is related to the systemic inflammation that underlies these conditions. Previous studies have shown that there are numerous types of immune cells in human adipose tissue, some of these are the macrophages. These cells can exist in two states: M2, which can inhibit classical inflammatory response, and M1 which secrete proinflammatory cytokines. The investigators have data to suggest that the role of inflammatory cells in adipose tissue is a strong contributor to systemic inflammation. A recent study showed that a GLP-1 analog (liraglutide, also known as Victoza) may help decrease inflammation via promoting M2 differentiation of macrophages. The purpose of this study is to quantify macrophage phenotype (M1 vs M2) in subcutaneous adipose tissue in moderately-obese diet controlled diabetics at baseline, after four weeks of weight-maintenance using liraglutide, and after 12 weeks of liraglutide treatment as compared to placebo.

Aim 1: Quantify M1 and M2 (surface and intracellular markers) polarization via flow cytometry in subcutaneous abdominal adipose tissue and peripheral blood mononuclear cells at baseline and after 4 weeks administration of liraglutide versus placebo to weight-stable, obese, type 2 diabetic patients. Weight loss will be prevented in order to ascertain the effect of liraglutide alone.

Aim 2: Quantify M1 and M2 (surface and intracellular markers) polarization via flow cytometry in subcutaneous adipose tissue and peripheral blood mononuclear cells after 12 weeks of liraglutide treatment, during which dietary restrictions are lifted and spontaneous weight loss, as would occur in the clinical setting, is allowed. To eliminate confounding by weight loss, a placebo-treated group will undergo matched dietary weight loss for comparison to the liraglutide group to ascertain whether changes in macrophage polarization at 12 weeks are greater in the liraglutide group.

Aim 3: Quantify macrophage-mediated localized and systemic inflammation by measuring M1/M2-related inflammatory cytokines in adipose tissue and peripheral blood after 4 and 12 weeks administration of liraglutide versus placebo to obese, type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 42 kg/m2
* Diet-controlled diabetics, or diabetics on Metformin that have permission from Primacy Care Physician to wash-out of the drug for 6 weeks prior to the study and for the duration of the study
* HbA1C between 6.0 - 7.9 (those on Metformin must have a HbA1c level below 7.5 prior to wash-out period)
* Fasting Blood Glucose < 150 mg/dl
* Women must be post-menopausal or surgically sterile within age range
* Subjects must live in vicinity of Stanford University

Exclusion Criteria:

* Prior Bariatric surgery
* Personal or family history of medullary thyroid cancer
* MEN2 Syndrome
* Thyroid Nodules (not evaluated by PCP)
* Pancreatitis (acute or chronic)
* Gallstones
* Fasting plasma triglycerides > 400 mg/dl
* Cardiovascular disease
* Major organ disease
* Unstable hypertension (BP >160/100 mm Hg)
* Heavy alcohol use
* Self-reported weight change of >2kg over past 6 weeks
* Medication known to affect blood glucose, insulin sensitivity, or inflammation
* NSAIDs (must cease use 4 weeks prior to study enrollment)
* Previous use of liraglutide, Januvia, Byetta, or Lira.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Macrophage polarization: % M2 macrophages in adipose tissue and peripheral blood according to positivity for cell surface markers (measured by flow cytometry). | 30 months

SECONDARY OUTCOMES:
Inflammation, localized: Pro- and anti-inflammatory cytokines will be measured (IL6, IL-8, TNF-α, MCP-1, cell surface markers, and adiponectin) by rtPCR in adipose tissue and blood macrophages | 30 months
Inflammation, systemic: Plasma pro/anti-inflammatory cytokines: IL-6, hsCRP, cell surface markers, and adiponectin will be measured in plasma. | 30 months
Macrophage polarization: M1 to M2 ratio in adipose tissue and peripheral blood according to cell surface markers (measured by flow cytometry) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University
Locations (1):
- Freidenrich Center for Translational Research (FCTR), Stanford, California, United States